CLINICAL TRIAL: NCT04500743
Title: Role of Suppression of Endometriosis With Progestins Before IVF-ET: a Non-inferiority Randomized Controlled Trial
Brief Title: Role of Suppression of Endometriosis With Progestins Before IVF-ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mazen Abdel Rasheed, Principal Investigator, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dienogest before IVF
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: IVF; Endometriosis; Pregnancy Rate; Progestins; GnRH-analogue
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Leuprolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dienogest (Active Comparator)
  Interventions: Drug: Dienogest
- GnRH analogue (Active Comparator)
  Interventions: Drug: leuprorelin acetate

INTERVENTIONS:
Drug: Dienogest — Group B (n=67) who had daily oral Dienogest 2 mg/d for 3 months before starting standard long protocol for IVF
  Arms: Dienogest
Drug: leuprorelin acetate — Group A (n=67) who had monthly depot GnRHa for 3 months before ovarian stimulation in IVF treatment (Ultra-long protocol)
  Arms: GnRH analogue

SUMMARY:
This study aimed to assess the role of Dienogest pretreatment for endometriosis suppression as compared to Gonadotropin-releasing hormone agonist (GnRHa) in patients with endometriosis pursuing IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of endometriosis
* body mass index < 35 Kg/m2

Exclusion Criteria:

* if they have been already on long-term down-regulation of the pituitary gland with GnRHa for control of endometriosis
* liver or kidney disease
* evidence of diminished ovarian reserve (e.g. high FSH level >12 IU/L or low AMH level <1 ng/ml).

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
the number of retrieved oocytes | After the ovarian induction (3 months after the pre treatment with either GnRHa or Dienogest)
  the number of retrieved oocytes as the main concern was the effect of either GnRHa or Dienogest on ovarian responsiveness

SECONDARY OUTCOMES:
the fertilization rate | After the ovarian induction (3 months after the pre treatment with either GnRHa or Dienogest)
  defined as the number of zygotes with two pronuclei divided by the number of oocytes
the number of transferrable embryos | After the ovarian induction (3 months after the pre treatment with either GnRHa or Dienogest)
  defined as the number of embryos suitable for transfer in the stimulated cycle or cryopreservation
the cost of the treatment | After the ovarian induction (3 months after the pre treatment with either GnRHa or Dienogest)
  the cost of the treatment in Egyptian pounds including cost of pretreatment and ovarian stimulation drugs
pregnancy rate per cycle started | After the ovarian induction (3 months after the pre treatment with either GnRHa or Dienogest)
  defined as patients with positive urinary or serum pregnancy test divided by the number of patients starting the treatment
the clinical pregnancy rate per cycle started | after women have postive pregnancy test (2 weeks after after the embryo transfer)
  defined as the number of patients with at least one intrauterine gestational sac with identifiable fetal heart pulsations over the total number of patients starting the treatment
the miscarriage rate | After occurence of the clinical pregnancy (5 months after after the embryo transfer)
  defined as patients with identified intrauterine gestational sac without a fetal pole, or a fetal pole with no heart pulsations with no other viable fetuses over the number of patients with positive pregnancy test
patient's quality of life | throughout the pre-treatment with GnRHa or Dienogest as well as the induction of ovulation "through study completion, an average of 9 months"
  patient's quality of life during the pretreatment period as assessed by the Fertility quality of life (FertiQoL) questionnaire with a range of 0 (the worst) to 100 (the best).

CONTACTS AND LOCATIONS:
Locations (1):
- Minia Infertility research unit, Minya, Egypt

REFERENCES:
- [Derived] Chen I, Kives S, Zakhari A, Nguyen DB, Goldberg HR, Choudhry AJ, Le AL, Kowalczewski E, Schroll JB. Progestagens for pain symptoms associated with endometriosis. Cochrane Database Syst Rev. 2025 Oct 9;10(10):CD002122. doi: 10.1002/14651858.CD002122.pub3. PMID 41065045
- [Derived] Khalifa E, Mohammad H, Abdullah A, Abdel-Rasheed M, Khairy M, Hosni M. Role of suppression of endometriosis with progestins before IVF-ET: a non-inferiority randomized controlled trial. BMC Pregnancy Childbirth. 2021 Mar 30;21(1):264. doi: 10.1186/s12884-021-03736-2. PMID 33784989